CLINICAL TRIAL: NCT06610864
Title: Surgical and Obstetric Outcomes in Patients With Uterine Malformations Undergoing Hysteroscopic Corrective Treatment
Acronym: MAL_CO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Catena Ursula, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6716
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-09

CONDITIONS: Malformation; Female Infertility; Hysteroscopy Surgery
Keywords: uterine malformation; hysteroscopic metroplasty; reproductive outcomes
MeSH Terms: conditions — Congenital Abnormalities; Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women with uterine malformations: Women with uterine malformations who underwent hysteroscopic correction.

SUMMARY:
The goal of this observational cohort study is to learn if hysteroscopic correction can improve reproductive outcomes in women with uterine malformations. The main questions it aims to answer are:

Primary hypothesis:

-Does hysteroscopic correction significantly improve pregnancy rates at 12 months post-surgery in women with uterine malformations?

Secondary hypotheses:

* Does hysteroscopic correction significantly reduce the rate of first and second-trimester spontaneous abortions?
* Does hysteroscopic correction significantly increase the live birth rate?
* In symptomatic patients, does hysteroscopic correction significantly reduce dyspareunia and dysmenorrhea?
* Which patient, histopathological, and surgical factors are associated with improved obstetric outcomes?

Researchers will compare obstetric outcomes (pregnancy rate, spontaneous abortion rate, live birth rate, and symptom severity) before and after hysteroscopic correction to determine the effectiveness of this surgical intervention.

Participants will be women with uterine malformations who underwent hysteroscopic correction at the Digital Hysteroscopy Center of Policlinico Universitario A. Gemelli di Roma and Azienda Ospedaliera Universitaria Federico II di Napoli. Data will be retrospectively collected and analyzed to assess the impact of surgery on reproductive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent hysteroscopy at the Class Hysteroscopy Center of Policlinico Universitario A. Gemelli di Roma or Azienda Ospedaliera Universitaria Federico II di Napoli for the correction of uterine malformations, including partial, complete, and septate bicornuate uteri, dysmorphic uteri, with or without associated cervical and/or vaginal septa (ESHRE-ESGE classification: U1a and U1c; U2a, U2b, and U3c with or without associated cervical or vaginal anomalies C1/2 or V1/2).
* Age 18 years or older.

Exclusion Criteria:

* Patients with known, concurrent causes of infertility.
* Patients who did not provide informed consent to participate in the study.
* Age younger than 18 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of women who underwent hysteroscopic correction for uterine malformations at the Class Hysteroscopy Center of Policlinico Universitario A. Gemelli di Roma or Azienda Ospedaliera Universitaria Federico II di Napoli. These malformations include partial, complete, and septate bicornuate uteri, dysmorphic uteri, with or without associated cervical and/or vaginal septa. Patients will be identified retrospectively through a review of medical records and will be contacted via telephone to obtain informed consent for participation in the study. Data will be collected retrospectively from medical records and through semi-annual follow-up telephone calls over a 12-month period.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-10-11 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rates | From January 2021 to December 2023
  To compare pregnancy rates (number of clinical pregnancies including live births, abortions and fetal deaths) before and after hysteroscopic correction in women with uterine malformations

SECONDARY OUTCOMES:
Abortion rate | From January 2021 to December 2023
  To compare rates of first and second-trimester spontaneous abortions before and after hysteroscopic correction
Live birth rate | From January 2021 to January 2023
  To compare live birth rates before and after hysteroscopic correction.
Symptoms resolution | From January 2021 to December 2023
  In a subgroup of symptomatic patients, to assess the impact of hysteroscopic correction on the reduction of dyspareunia and dysmenorrhea
Prognostic factors | From January 2021 to December 2023
  To identify potential prognostic factors, including medical history, histopathology, and surgical factors, associated with improved obstetric outcomes following hysteroscopic correction.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Catena, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrera M, Perez Millan F, Alcazar JL, Alonso L, Caballero M, Carugno J, Dominguez JA, Moratalla E. Effect of Hysteroscopic Metroplasty on Reproductive Outcomes in Women with Septate Uterus: Systematic Review and Meta-Analysis. J Minim Invasive Gynecol. 2022 Apr;29(4):465-475. doi: 10.1016/j.jmig.2021.10.001. Epub 2021 Oct 11. PMID 34648934
- [Background] Grimbizis GF, Camus M, Tarlatzis BC, Bontis JN, Devroey P. Clinical implications of uterine malformations and hysteroscopic treatment results. Hum Reprod Update. 2001 Mar-Apr;7(2):161-74. doi: 10.1093/humupd/7.2.161. PMID 11284660